CLINICAL TRIAL: NCT06990126
Title: A Real World Study on the Clinical Efficacy and Adverse Reactions of Neotetracycline Drugs in the Treatment of Gram-negative Bacterial Infections
Brief Title: The Efficacy and Adverse Reactions of Neotetracycline in the Treatment of GNB Infections
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-SR-268
Record Dates: First submitted 2025-04-17; First posted 2025-05-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-05

CONDITIONS: Clinical Efficacy and Safety
Keywords: Eravacycline; Tigecycline; Gram-negative bacteria; adverse drug reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Bronchoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: bronchoscope — We will perform bronchoscopy and collect bronchoalveolar lavage fluid(BALF)

SUMMARY:
A multicenter, retrospective, real-world stduy . Subjects with composite criteria were teated with eravacycline ,and 100 cases ,Tigecycline and 300 cases were to be enrolled.

DETAILED DESCRIPTION:
The study is a multicenter, retrospective, real-world study, through retrospective collection of cases of gram-negative bacterial infections in the First Affiliated Hospital of Nanjing Medical University, Nanjing Drum Tower Hospital, Nanjing First Hospital, Shaw Hospital Affiliated to Nanjing Medical University, Affiliated Hospital of Xuzhou Medical University, and Xuzhou Central Hospital, and 100 cases of eravacycline,300 cases of tigecycline are planned to be enrolled.

Inclusion Criteria:

Bacteriological results show drug-resistant Gram-negative bacteria Use of new tetracycline drugs for ≥72 hours Age ≥18 years

Exclusion Criteria:

Advanced tumors Severe immunodeficiency or mental illness Severe liver and kidney dysfunction Pregnant or breastfeeding women Rejection Criteria: None

Data acquisition:

General condition: age, gender, acute physiology and chronic health status score (APACHEII), endotracheal intubation/tracheostomy, site of infection, course of treatment, presence of other pathogens, concomitant use of other antibiotics, and ICU admission; Specimen source: blood/respiratory/other; Drug-resistant pathogens: Acinetobacter baumannii/Klebsiella pneumoniae/Escherichia coli; Evaluation of clinical efficacy and bacterial efficacy during treatment with eravacycline and tigecycline; Common adverse reactions in eravacycline or tigecycline therapy; Treatment options Recommended dose of eravacycline : calculated according to the patient's weight, intravenous infusion at 1mg/kg, q12h, the infusion duration is not less than 60 minutes, and the recommended course of treatment is 4-14 days. The investigator can adjust the specific medication regimen according to the severity and location of the patient's infection and the patient's clinical response.

Recommended dose of tigecycline is 100 mg as a loading dose and 50 mg every 12 hours as a maintenance dose, and for multidrug-resistant infections, a high-dose tigecycline 200 mg as an initial dose and a maintenance dose up to 100 mg every 12 hours.

ELIGIBILITY:
Inclusion Criteria:

Bacteriological results show drug-resistant Gram-negative bacteria Use of new tetracycline drugs for ≥72 hours Age ≥18 years

Exclusion Criteria:

Advanced tumors Severe immunodeficiency or mental illness Severe liver and kidney dysfunction Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infections clinically caused by drug-resistant gram-negative bacteria (other than CRPA) and treated with eravacycline and tigecycline
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 14 days
  The main outcome is the clinical results of assessed by clinical physicians, where clinical outcomes are recorded as successful or unsuccessful, defined by the relief of clinical symptoms, which is defined as imaging improvement determined by the clinician, normalization or significant reduction of white blood cell counts and related inflammatory indicators including CRP, PCT, IL-6, etc.

SECONDARY OUTCOMES:
Microbiological efficacy and safety | 14 days
  The secondary outcome is the microbiological efficacy, namely the control of bacterial infections during hospitalization (including the clearance and partial clearance of bacteria) and safety, which is assessed by evaluating the incidence of adverse events and changes in clinical laboratory test results (including liver and kidney functions, coagulation function, etc.) for all study subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China